CLINICAL TRIAL: NCT06213831
Title: A Maximal Use Trial of Ruxolitinib Cream in Adult Participants With Prurigo Nodularis
Brief Title: A Study to Evaluate the Safety and Tolerability of Maximal Use Ruxolitinib Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB18424-110
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo Nodularis; PN; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Maximal Use Ruxolitinib 1.5% (Experimental): Participants will apply ruxolitinib 1.5% cream BID through Week 4 to all pruriginous lesions. At Week 4, participants who have completed 4 weeks of treatment with no safety concerns may enter the optional 4-week treatment extension period, during which all participants will apply ruxolitinib 1.5% cream BID to existing pruriginous lesions.
  Interventions: Drug: Ruxolitinib Cream 1.5%

INTERVENTIONS:
Drug: Ruxolitinib Cream 1.5% — Ruxolitinib Cream 1.5%

SUMMARY:
This study is being conducted to determine the safety and tolerability of ruxolitinib 1.5% cream under maximal use conditions in participants with Prurigo Nodularis (PN).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PN ≥ 3 months before screening.
* Pruriginous lesions (defined as papules, nodules, plaques, umbilicated lesions, and linear lesions) on ≥ 2 different body areas (such as right and left leg) at screening and baseline.
* Total estimated treatment BSA ≥ 25% (excluding the scalp) at screening and baseline.
* IGA-CPG-S score of ≥ 2 at screening and baseline.
* Baseline PN-related WI-NRS score ≥ 7. Baseline WI-NRS score is defined as the 7-day average of WI-NRS scores before Day 1 (data from a minimum of 4 out of 7 days prior to Day 1 is needed).

Exclusion Criteria:

* Chronic or acute pruritus due to a condition other than PN.
* Active AD lesions (signs and symptoms other than dry skin) within 6 months of screening and baseline.
* Acute or chronic active HBV or HCV infection.
* Any underlying condition known to be associated with the clinical presentation of PN that is not under control (stable) prior to the baseline visit.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 16 weeks, including 30 days of safety follow-up
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Number of participants with TEAEs leading to dose interruption or discontinuation | Up to 16 weeks, including 30 days of safety follow-up
  Number of participants with TEAEs leading to dose interruption or discontinuation.

SECONDARY OUTCOMES:
Ruxolitinib pharmacokinetic (PK) parameters in plasma | Up to 16 weeks, including 30 days of safety follow-up
  Ruxolitinib concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (20):
- United States (20):
  - Saguaro Dermatology, Phoenix, Arizona
  - Affiliated Dermatology, Scottsdale, Arizona
  - First Oc Dermatology, Fountain Valley, California
  - Amicis Research Center Valencia, Northridge, California
  - Clinical Science Institute Clinical Research Specialists Inc, Santa Monica, California
  - Advanced Pharma Cr, Llc, Miami, Florida
  - Sullivan Dermatology North Miami Beach Office, North Miami Beach, Florida
  - Olympian Clinical Research, Tampa, Florida
  - St Lukes Clinic Dermatology Ketchum, Ketchum, Idaho
  - Dawes Fretzin Clinical Research Group Llc, Indianapolis, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - Oakland Hills Dermatology Pc, Auburn Hills, Michigan
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Equity Medical, Llc, New York, New York
  - Red River Research Partners, Fargo, North Dakota
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Paddington Testing Co Inc, Philadelphia, Pennsylvania
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Dermresearch, Inc., Austin, Texas
  - North Texas Center For Clinical Research Ntccr, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study to evaluate the safety and tolerability of maximal use Ruxolitinib Cream — https://www.incyteclinicaltrials.com/study/?id=INCB18424-110&SearchTerm=INCB18424-110&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=